CLINICAL TRIAL: NCT00139711
Title: A Multicenter Randomized Phase II Study Evaluating The Activity And Tolerability Of Three Different Combinations Of Docetaxel (Taxotere) And Irinotecan (Campto) As Second Line Therapy For Recurrent Or Metastatic Non Small Cell Lung Cancer (NSCLS)
Brief Title: Three Combinations Of Docetaxel And Irinotecan For Recurrent Or Metastatic Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976C/2501; A5961088
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2006-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Irinotecan; Docetaxel

INTERVENTIONS:
Drug: Irinotecan
Drug: Docetaxel

SUMMARY:
A multicenter randomized phase II study evaluating the activity and tolerability of three different combinations of docetaxel (taxotere) and irinotecan (campto) as second line therapy for recurrent or metastatic non small cell lung cancer (NSCLC)

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven NSCLC
* Recurrent or metastatic NCSLC

Exclusion Criteria:

* Prior malignancies; except for cured non melanoma skin cancer, curatively treated in situ carcinoma of the cervix or other cancer adequately treated an with non evidence of disease for at least 5 years
* History or presence of brain or meningeal metastases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138
Dates: Start 2003-03; Study Completion 2006-06

PRIMARY OUTCOMES:
Evaluate the activity and tolerability of the association of irinotecan and docetaxel according to three different schedules as second line treatment for recurrent or metastatic NSCLC.

SECONDARY OUTCOMES:
Evaluate, in each arm, the time to progression, the duration of response and the survival

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- Italy (15):
  - Pfizer Investigational Site, Alzano Lombardo, BG
  - Pfizer Investigational Site, Gravedona, CO
  - Pfizer Investigational Site, Crema, CR
  - Pfizer Investigational Site, Gorgonzola, MI
  - Pfizer Investigational Site, Melegnano, MI
  - Pfizer Investigational Site, Vimercate, MI
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Benevento
  - Pfizer Investigational Site, Borgomanero
  - Pfizer Investigational Site, Brescia
  - Pfizer Investigational Site, Mantova
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Monza
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Varses

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=XRP6976C/2501&StudyName=Three+Combinations+Of+Docetaxel+And+Irinotecan+For+Recurrent+Or+Metastatic+Non+Small+Cell+Lung+Cancer+